CLINICAL TRIAL: NCT01753505
Title: Clinical Significance of 64-slice Multidetector Coronary CT Angiography to Evaluate the Prevalence and Severity of Coronary Artery Disease in Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4-2012-0549
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Kidney Transplant Recipient
Keywords: multidetector coronary CT angiography, renal transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDCTA (Experimental)
  Interventions: Other: 64-slice Multidetector coronary CT angiography

INTERVENTIONS:
Other: 64-slice Multidetector coronary CT angiography

SUMMARY:
The aim of this study is to evaluate the clinical usefulness of 64-slice multidetector coronary CT angiography (MDCTA) in renal transplant recipients who had no previous coronary artery disease (CAD). Primary endpoint is to assess the prevalence and severity of coronary artery disease in patients post-transplant 6 to 12 months. CAD can be diagnosed noninvasively with similar accuracy of coronary angiography using MDCTA. Early detection and intervention of CAD may provide survival benefit in renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 40 yrs
2. renal transplant recipient at post-transplant 6 to 12 months
3. stable graft renal function: CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) equation ≥45 mL/min/1.75m2
4. patients who had no previous CAD

Exclusion Criteria:

1. unstable graft renal function
2. History of acute kidney injury within 3 months
3. Allergic history to contrast agent
4. Irregular heart beat
5. Multiorgan transplant recipients
6. Pregnancy
7. Patients who do not consent to this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2014-07-28 (Actual); Study Completion 2014-07-28 (Actual)

PRIMARY OUTCOMES:
prevalence of coronary artery disease | at post-transplant 6 to 12 months.

SECONDARY OUTCOMES:
severity of coronary artery disease | at post-transplant 6 to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea